CLINICAL TRIAL: NCT01651897
Title: Delirium in the Emergency Department and Its Extension Into Hospitalization
Acronym: DELINEATE
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jin H. Han, MD, MSc, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 111580
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Delirium
Keywords: delirium; emergency department; natural course; outcomes; elderly
MeSH Terms: conditions — Delirium; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 15-30 cc of blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delirious in the ED: Patients who were delirious in the ED at either the 0-hour or 3-hour delirium assessment.
- Non-Delirious in the ED: Patients who were non-delirious in the ED at both the 0-hour or 3-hour delirium assessment.

SUMMARY:
Delirium occurs in 10% of older emergency department (ED) patients, yet it remains poorly understood. To date, the predominance of delirium studies have been conducted in hospitalized patients and therefore have limited generalizability to the ED. Understanding ED delirium's natural course and its effect on outcomes is not well characterized. The investigators hypothesize that a significant proportion of patients who are delirious in the ED will remain delirious in the hospital, and persistent cases of ED delirium will be significantly associated with higher 6-month mortality and accelerated functional decline. To test this hypothesis, the investigators will perform a prospective cohort study that will enroll 150 older ED patients with delirium and a random selection of 150 older ED patients without delirium; both groups will comprise of admitted ED patients only. Once enrolled in the ED, the investigators will assess patients for 7 days during hospitalization and perform phone follow-up at 6-months.

DETAILED DESCRIPTION:
Delirium is an acute confusional state characterized by fluctuating mental status, inattention, and either disorganized thinking or an altered level of consciousness. The prevalence of delirium in elderly patients is approximately 10% in emergency department (ED) patients. Several hospital-based studies have shown delirium to be associated with worsening mortality,longer hospital length of stay, higher health care costs,and poorer long-term functional and cognitive function.

However, delirium in the ED remains poorly understood. Specifically, its natural course is not well characterized and represents a critical gap in knowledge. Improving our understanding is paramount for several reasons. If the majority of delirium persists beyond the ED and is associated with long-term adverse outcomes, then routine delirium surveillance in the busy ED environment can be justified. Understanding the natural course may also help physicians identify delirious patients at highest risk for adverse outcomes and would be the focus of future delirium interventions. Lastly, we don't know if all patients with delirium require an admission. Understanding the natural course may help identify delirious patients that can be safely discharged home and those who require a hospital admission.

Given this paucity of data, we are conducting this study with the following specific aims: 1) To describe the frequency in which delirium in the ED persists into hospitalization and determine how patient factors and clinical factors affect delirium persistence. 2) To determine how ED delirium duration affects 6-month outcomes. To achieve these aims, we will perform a prospective cohort study thatwill enroll 125 older ED patients with delirium and a random selection of 125 older ED patients without delirium; both groups will comprise of admitted ED patients only. Once enrolled in the ED, we will assess patients for 7 days during hospitalization and perform phone follow-up at 6-months.

ELIGIBILITY:
Inclusion Criteria:

* 65 Years and older
* In an ED bed for less than 4 hours at the time of enrollment
* Any possibility of being admitted to the hospital

Exclusion Criteria:

* Refuse consent
* Have been previously enrolled
* Unarousable to verbal stimuli
* Have severe mental retardation or severe dementia characterized by being non-verbal or unable to comprehend simple instructions at baseline
* Deaf
* Patient or surrogate is non-English speaking
* Discharged from the emergency department

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will enroll 150 delirious ED patients and a random selection of 150 non-delirious ED patients who are hospitalized and reassess their delirium status daily throughout their hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
6-month mortality and functional status. | 6-months
  We will perform 6-month phone follow-up to ascertain death and functional status.
Emergency department delirium duration | Until hospital discharge or the first 7-days of hospitalization.
  Patients will be enrolled in the emergency department and will be assessed for delirium daily until hospital day #7 or hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States